CLINICAL TRIAL: NCT05985070
Title: Evaluating the Effectiveness of Various Iron Salts in Oral Iron Therapy for Iron Deficiency and Anemia in Healthy Adults: A Multicenter, Randomized, Double-blind, Parallel-group Pragmatic Clinical Trial
Brief Title: Evaluating the Effectiveness of Various Iron Salts in Oral Iron Therapy for Iron Deficiency and Anemia in Healthy Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liaquat University of Medical & Health Sciences (Other)
Responsible Party: Principal Investigator, Dr. Nazia Mumtaz Memon, Assistant Professor Pathology, Liaquat University of Medical & Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LUMHS/REC/-86
Record Dates: First submitted 2023-08-02; First posted 2023-08-14 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-04

CONDITIONS: Iron Deficiency; Iron Deficiency Anemia
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency | interventions — sucrosomial iron; ferric maltol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm 1 (Experimental): Subjects in this arm will receive an oral Sucrosomial 30mg elemental iron supplement, twice daily, for 6 weeks.
  Interventions: Dietary Supplement: Oral Sucrosomial iron
- Intervention Arm 2 (Active Comparator): Subjects in this arm will receive an oral Ferric maltol 30mg elemental iron supplement, twice daily, for 6 weeks.
  Interventions: Dietary Supplement: Oral Ferric maltol

INTERVENTIONS:
Dietary Supplement: Oral Sucrosomial iron — 30 mg capsule
  Arms: Intervention Arm 1
Dietary Supplement: Oral Ferric maltol — 30 mg capsule
  Arms: Intervention Arm 2

SUMMARY:
Oral iron supplements are a cornerstone therapy for treating iron deficiency and iron deficiency anemia, aiming to replenish low iron levels in the body. These supplements typically contain various iron salts, such as ferrous sulfate, ferric maltol, ferrous gluconate, and ferric pyrophosphate.

Advancements in carrier systems, such as microencapsulation or complexation can enhance the absorption and bioavailability of iron supplements. By improving absorption, these carrier systems may mitigate gastrointestinal side effects and increase the efficacy of iron therapy.

DETAILED DESCRIPTION:
This multicenter, randomized, double-blind parallel-group, clinical trial study aims to conduct a comparative analysis of the effectiveness of oral ferric maltose, vs Sucrosomial iron. The study seeks to evaluate their efficacy in treating iron deficiency or iron deficiency anemia, two prevalent conditions associated with low iron levels in the body. This research aims to provide valuable insights into potential difference in these two iron supplement formulations, both in terms of relative effectiveness and potential GI side effects. This comparative analysis may guide healthcare providers in selecting the most suitable oral iron supplement based on individual patient characteristics, ultimately optimizing treatment outcomes and improving patient care.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adults aged 18-65 years
* Iron deficiency, defined as low serum iron <50 µg/dL, ferritin <20 ng/mL, and TIBC >400 µg/dL.
* Able and willing to provide informed consent
* Willing to comply with oral supplementation and study follow-up

Exclusion Criteria:

* Severe anemia, defined as hemoglobin (Hb) <8 g/dL, requiring urgent intervention
* Known malabsorption syndromes (e.g., celiac disease, IBD)
* Active bleeding or blood transfusion within the past 3 months
* Pregnancy or lactation
* Use of iron supplements within the past 4 weeks
* Known allergy or intolerance to oral iron formulations

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the serum iron concentration | 6 weeks
  Increase in the circulatory iron levels
Changes in the serum ferritin concentration | 6 weeks
  Increase in the circulatory ferritin levels
Change in blood Hemoglobin (Hb) levels | 6 weeks
  Increase in the blood (Hb) levels

OTHER OUTCOMES:
Incidence of gastrointestinal side effects | 6 weeks
  Incidence of treatment-emergent gastrointestinal side effects

CONTACTS AND LOCATIONS:
Locations (3):
- Pakistan (3):
  - Mayo Hospital, Lahore, Punjab Province
  - DHQ Hospital Narowal, Narowal, Punjab Province
  - Civil Hospital Kotri Distt Jamshoro, Kotri, Sindh

IPD SHARING:
Plan to Share IPD: No